CLINICAL TRIAL: NCT01767688
Title: An Open-Label, Single-Dose Study to Investigate the Pharmacokinetics of MK-3102 in Patients With Impaired Hepatic Function
Brief Title: A Pharmacokinetic Study of MK-3102 in Participants With Impaired Hepatic Function (MK-3102-031)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3102-031
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Hepatic Impairment Group (Experimental)
  Interventions: Drug: MK-3102
- Healthy Matched Control Group (Experimental)
  Interventions: Drug: MK-3102

INTERVENTIONS:
Drug: MK-3102 — Single dose of 25 mg of MK-3102 (1 x 25 mg capsule) administered orally on Day 1.

SUMMARY:
This study will investigate and compare the pharmacokinetics of a single 25-mg dose of MK-3102 in participants with moderate hepatic impairment and matched healthy participants. The primary hypothesis is that in participants with moderately impaired hepatic function, the area under the concentration-time curve from time zero to infinity (AUC0-∞) is similar to that observed in healthy matched control participants following a single 25 mg oral dose of MK-3102. Specifically, the true ratio (moderately impaired hepatic function patients/healthy matched control subjects) of geometric means for AUC0-∞ is no greater than 2.

ELIGIBILITY:
Inclusion Criteria:

Impaired Hepatic Function Participants:

* A diagnosis of:

  1. Chronic (> 6 months) hepatic insufficiency
  2. Stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology
* Score on the Child-Pugh Scale of 7 to 9 (moderate hepatic insufficiency)
* Estimated creatinine clearance (CLCr) > 60 mL/min or glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m^2

Both Impaired Hepatic Function and Healthy Participants:

* In general good health
* Continuous non-smokers or moderate smokers for at least 3 months prior to study start
* Body Mass Index ≤39 kg/m^2
* Females of reproductive potential must have a negative pregnancy test and agree to use acceptable birth control method(s) or remain sexually inactive throughout study
* Non-vasectomized male patients must agree to use acceptable birth control method(s) or abstain from sexual intercourse during the trial and for 3 months after the study

Exclusion Criteria:

Healthy Participants:

* History or presence of alcoholism within the past 2 years
* Presence of hepatitis B virus (HBV) or hepatitis virus C (HVC)

Both Impaired Hepatic Function and Healthy Participants:

* History or presence of drug abuse within the past 2 years
* History or presence of human immunodeficiency virus (HIV)
* History or presence of significant cardiovascular, pulmonary, renal, hematologic, gastrointestinal (other than hepatic impairment), endocrine, immunologic, dermatologic, or neurological disease
* Use of any medication or substance (including prescription or over the counter, health supplements, natural or herbal supplements) which cannot be

discontinued at least 14 days prior to the study start and throughout the study

* Has been on a special diet within 28 days prior to the study start
* Blood donation within 56 days or plasma donation within 7 days prior to study start
* Participation in another clinical trial within 28 days of study start
* Women who are pregnant or nursing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-07 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=3102-031&kw=3102-031&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult (18 to 80 years of age) males and females participated in the study. Eight participants with moderate hepatic impairment, and eight healthy control participants (matched according to age, weight, gender, and creatinine clearance [CLCr] or estimated glomerular filtration rate [eGFR]), were enrolled.
Groups:
- Moderate Hepatic Impairment Group: Participants with Child-Pugh scores of 7-9 were enrolled in the Moderate Hepatic Impairment group.
- Healthy Matched Control Group: Healthy participants matched according to mean age (±15 years), mean weight (±10 kg), and mean CLCr (±20 mL/min) or mean eGFR (±20 mL/min/1.73 m²) to same-gender participants with moderate hepatic impairment were enrolled in the Control group.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: Years] | 57 (6.45) [45 to 62] | 53 (8.45) [41 to 68] | 55 (7.55) [41 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Hour 0 to Infinity (AUC0-∞)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 96, and 168 hours post-dose
Population: All participants that received omarigliptin 25 mg.
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
µM*hr | 23.3 [20.2 to 26.9] | 24.9 [21.8 to 28.3]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Healthy Matched Control Group; Test type: Superiority or Other; Geometric least-squares mean ratio (GMR); Geometric least-squares mean ratio (GMR) = 0.94, 95% CI 2-sided [0.79 to 1.11]

2. Secondary Outcome: Area Under the Concentration Versus Time Curve From Hour 0 to 168 Hours After Dosing (AUC0-168h)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 96, and 168 hours post-dose
Population: All participants that received omarigliptin 25 mg.
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
µM*hr | 22.4 [19.8 to 25.4] | 23.8 [21.2 to 26.7]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Healthy Matched Control Group; Test type: Superiority or Other; Geometric least-squares mean ratio (GMR); Geometric least-squares mean ratio (GMR) = 0.94, 95% CI 2-sided [0.81 to 1.10]

3. Secondary Outcome: Plasma Concentration at 168 Hours After Dosing (C168h)
Time Frame: 168 hours post-dose
Population: All participants that received omarigliptin 25 mg.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
nM | 15.7 [10.7 to 23.0] | 19.4 [13.7 to 27.4]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Healthy Matched Control Group; Test type: Superiority or Other; Geometric least-squares mean ratio (GMR); Geometric least-squares mean ratio (GMR) = 0.81, 95% CI 2-sided [0.51 to 1.28]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 96, and 168 hours post-dose
Population: All participants that received omarigliptin 25 mg.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
nM | 572 [523 to 626] | 554 [511 to 600]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment Group vs Healthy Matched Control Group; Test type: Superiority or Other; Geometric least-squares mean ratio (GMR); Geometric least-squares mean ratio (GMR) = 1.03, 95% CI 2-sided [0.93 to 1.15]

5. Secondary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 96, and 168 hours post-dose
Population: All participants that received omarigliptin 25 mg.
Measure: Median (Full Range); unit: hr
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
hr | 2 [1 to 4] | 2 [2 to 4]

6. Secondary Outcome: Apparent Terminal Phase Half-life (t½)
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 96, and 168 hours post-dose
Population: All participants that received omarigliptin 25 mg.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
hr | 34.6 (17.4) | 34.5 (13.4)

7. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation patient/subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 14 days post-dose
Population: All participants that received omarigliptin 25 mg.
Measure: Number; unit: Participants
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
Participants | 2 | 1

8. Secondary Outcome: Number of Participants Discontinued From Study Due to AEs
Description: as for outcome 7
Time Frame: Up to 14 days post-dose
Population: All participants that received omarigliptin 25 mg.
Measure: Number; unit: Participants
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were monitored for 14 days after receiving omarigliptin 25 mg.
Arm/Group | Moderate Hepatic Impairment Group | Healthy Matched Control Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Impairment Group (N=8) | Healthy Matched Control Group (N=8)
Headache (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will provide separate guidance on the criteria for publication of clinical trial data when contacted for permission to publish.